CLINICAL TRIAL: NCT04158700
Title: Phase 1b/2 Study of LY3200882 and Pembrolizumab in Patients With Advanced Cancer
Brief Title: A Study of LY3200882 and Pembrolizumab in Participants With Advanced Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The withdrawal is due to a strategic realignment and is not related to any particular safety or efficacy concern.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17387; I8X-MC-JECD (Other: Eli Lilly and Company); 2019-001156-18 (EudraCT Number); KEYNOTE-961 (Other: Merck)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Advanced Cancer
Keywords: TGF-beta; Urothelial carcinoma; Hepatocellular carcinoma; Non-small cell lung cancer; TGF- beta receptor type I inhibitor
MeSH Terms: conditions — Camurati-Engelmann Syndrome; Carcinoma, Transitional Cell; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3200882 and Pembrolizumab (Dose Level 1) (Experimental): Participants with urothelial carcinoma: LY3200882 administered orally with pembrolizumab administered intravenously (IV).
  Interventions: Drug: LY3200882; Drug: Pembrolizumab
- LY3200882 and Pembrolizumab (Dose Level 2) (Experimental): Participants with urothelial carcinoma: LY3200882 administered orally with pembrolizumab administered IV.
  Interventions: Drug: LY3200882; Drug: Pembrolizumab
- LY3200882 and Pembrolizumab Expansion (Experimental): Participants with urothelial carcinoma, non-small cell lung cancer, or hepatocellular carcinoma: LY3200882 administered orally twice in combination with pembrolizumab administered IV.
  Interventions: Drug: LY3200882; Drug: Pembrolizumab

INTERVENTIONS:
Drug: LY3200882 — LY3200882 administered orally
Drug: Pembrolizumab — Pembrolizumab administered IV

SUMMARY:
The main purpose of this study is to see if the drug LY3200882 which is an inhibitor of transforming growth factor-β (TGFβ) receptor 1 in combination with pembrolizumab is safe and effective in participants with cancer that has spread to other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have received a PD-1 PDLI therapy within 9 weeks of starting dosing on this study [for example, nivolumab, pembrolizumab, atezolizumab]
* Participants must be willing to have tumor biopsies
* Participants must have adequate organ function
* Participants must have Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Participants must be able to swallow tablets
* Participants with stable, previously treated brain metastases may participate if neurologic symptoms have resolved and participants have been off steroids for at least 14 days

Exclusion Criteria:

* Participants must not have moderate or severe cardiovascular disease
* Participants must not have active autoimmune disease (for example Crohn's disease, Hashimotos disease, etc)
* Participants must not have an active infection requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-05 (Estimated); Primary Completion 2023-05-11 (Estimated); Study Completion 2023-05-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) | Up to 6 Weeks
  Number of Participants with DLT

SECONDARY OUTCOMES:
Overall Response Rate (ORR): Percentage of Participants with Complete Response (CR) or Partial Response (PR) | Baseline through Disease Progression or Death (Estimated at up to 12 Months)
  ORR: Percentage of Participants with CR or PR
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3200882 in Combination With Pembrolizumab | Baseline through Week 13
  PK: Cmax of LY3200882 in Combination With Pembrolizumab
Duration of Response (DoR) | Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (Estimated at up to 12 Months)
  DoR

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States
- France (2):
  - CHU de Besancon Hopital Jean Minjoz, Besançon
  - Gustave Roussy, Villejuif
- Spain (3):
  - Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Madrid Norte Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3200882 and Pembrolizumab in Participants With Advanced Cancer — https://www.lillytrialguide.com/en-US/studies/advanced-cancer/JECD#?postal=